CLINICAL TRIAL: NCT06709664
Title: Experiences of the Perimenopause and Menopause in Women With Spinal Cord Injury
Brief Title: Perimenopause and Menopause in Women With Spinal Cord Injury
Status: Not yet recruiting | Type: Observational
Sponsor: James Cooper (Other)
Responsible Party: Sponsor-Investigator, James Cooper, Research and Innovation Manager/Sponsor Representative, Buckinghamshire Healthcare NHS Trust
Organization: Buckinghamshire Healthcare NHS Trust (Other)
Other Study IDs: RXQ 1192
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Menopause; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with Spinal Cord Injury: Women with Spinal Cord Injury who are currently going through or have gone through the Perimenopause/Menopause
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire study

SUMMARY:
A lot of information is known about how the perimenopause and menopause affects able bodied women. However there is very little information about how these affects women with spinal cord injury. This questionnaire study aims to collect information from women with a spinal cord injury on their experiences of going through the perimenopause and/or the menopause.

DETAILED DESCRIPTION:
There is widespread knowledge and information about the perimenopause and menopause, its symptoms and treatment; all of this is for people without spinal cord injury (women will be used to denote all people who can or have undergone the perimenopause and menopause). There is paucity of data about this condition in women with spinal cord injury. These women are living longer lives and should be supported to live a healthy life.

Some studies have suggested that women with Spinal Cord Injury (wSCI) may undergo the perimenopause and menopause earlier than those without, however others have concluded that the age at the perimenopause and menopause is no different. wSCI may suffer less with vasomotor symptoms due to their ability to manage the symptoms of autonomic dysreflexia; however they may have more genito-urinary symptoms; also due to the need for self-catheterisation.

Hormone Replacement Therapy (HRT) has many benefits including reduction in risk of fractures by slowing down the development of osteoporosis, thereby reducing fracture risk and morbidity. Reduced mobility also puts them at an increased risk of cardio-vascular disease.

This study aims to gain information about these characteristics of the perimenopause and menopause in wSCI; the age at which they become menopausal and the most bothersome symptoms for them, treatment options offered to them as well as details of their spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* • Patient is willing and able to give informed consent for participation in the study (or verbally confirm they wish to take part if someone completing on their behalf)

  * Who has undergone or currently experiencing the perimenopause or menopause
  * Aged 18 years old or older
  * Clinically diagnosed with a spinal cord Injury at least 3 months ago
  * Is either a) currently going through the perimenopause and menopause or b) has been through the perimenopause and menopause.

Exclusion Criteria:

* • Individuals who have yet to go through the perimenopause and/or menopause

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women will be used to denote all people who can or have undergone the perimenopause and menopause
Study Population: women will be used to denote all people who can or have undergone the perimenopause and menopause and have a clinical diagnosis of a spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To collect more information on determine signs, symptoms and severity of these signs and symptoms of the perimenopause and menopause in women with spinal cord injury | 1 time point
  * Information on menstrual cycle
  * Frequency of autonomic dysreflexia
  * Typical signs of autonomic dysreflexia
  * Menopausal symptoms
  * Treatment for menopausal symptoms
  * Satisfaction of medication (for menopausal symptoms)
  * Satisfaction of support for the perimenopause and menopause

SECONDARY OUTCOMES:
To collect more information on establish how SCI affects the experience of the perimenopause and menopause | 1 time point
  * Patterns between level of injury and the perimenopause and menopause symptoms
  * Patterns between neurological level and the perimenopause and menopause symptoms

IPD SHARING:
Plan to Share IPD: Undecided